CLINICAL TRIAL: NCT03640806
Title: QOL Efficacy of Adapted Physical Activity for Patients With Fibromyalgia : Single-center, Prospective, Randomized With Biological and Cerebral Evaluation
Brief Title: QOL Efficacy of Adapted Physical Activity for Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-57
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHYSICAL ACTIVITY (Experimental): Standard support for 12 months (HAS 2010, EULAR 2016) 3 fibromyactiv workshops per week during the first 6 months, or 72 sessions. Each workshop lasts 2 hours of physical activity.
  Interventions: Other: PHYSICAL ACTIVITY
- CONTROL (No Intervention): Standard care for 12 months (HAS 2010, EULAR 2016) with Pain Consultation every 3 months.

INTERVENTIONS:
Other: PHYSICAL ACTIVITY — 3 fibromyactiv workshops per week during the first 6 months, or 72 sessions. Each workshop lasts 2 hours of physical activity.
  Arms: PHYSICAL ACTIVITY

SUMMARY:
Fibromyalgia affects at least 4% of the population. This chronic painful pathology is a source of social exclusion with a major impact on professional activity;

To our knowledge, no study has demonstrated with sufficient evidence the effectiveness of the practice of well-defined adapted physical activity (APA) via a reproducible program of physical activity that has been the mechanisms of action that underlie this efficacy by biology and functional brain imaging (PET CT) in this context.

In addition, the publications mention recruitment difficulties, a high drop-out rate and a difficult maintenance of the benefits of physical activity in the long term, or even a return to the initial level after a few months.

The programs evaluated do not seem to take into account the peculiarities of patients, their coping coping strategies, associated with chronic pain and disability . In order to reinforce the durability of the benefits of our intervention, we make modulating factors of "coping" styles of therapeutic targets in their own right, as well as muscular strength, aerobic capacity or flexibility. Thus, cognitive-behavioral therapy (CBT) procedures validated in the treatment of chronic pain are adapted and transposed to our APA program in order to propose specific strategies.

"Fibromy'activ" aims to act upstream and downstream of the formation of health inequalities found in the population suffering from fibromyalgia and favored by the natural evolution of the disease: These workshops tend to favorably influence the course of life and to define a reproducible interdisciplinary protocol.

It is a question of making accessible and reproducible the practice of adapted physical activity (APA), non-medicinal therapeutic recommended by the HAS since 2010 , by the EULAR in 2016, but not refunded, poorly protocolized therefore not reproducible and little implementation. It is part of the spirit of the amended Health Act with the coming into force of the application decree since March 2017 "Physical Prescription".

DETAILED DESCRIPTION:
Fibromy'activ, an adapted physical activity program (APA) for patients with fibromyalgia, aims to provide lasting symptomatic relief, to favorably influence the life course, to identify mechanisms of action and to define a reproducible interdisciplinary protocol.

Fibromyalgia affects at least 4% of the population. This chronic painful pathology is a source of social exclusion with a major impact on professional activity . In France, the prevalence of co-morbidities is increased in pain patients . There is a significant impact on health care systems. It is very expensive for the society of about € 7,900 / patient / year.

The fibromyalgia population managed at the Center for Assessment and Treatment of Pain CHU Timone (CETD), is characterized as follows: 50 years of average age, 85% of women with children in 80% of cases. 60% have a level of education lower than the baccalaureate, less than 30% have a professional activity. The duration of the pain before the first consultation is on average 8.1 years. The SPICE score is above average which indicates a higher level of precariousness. It is associated with dysfunctional pain adjustment strategies, psychological distress, low acceptance and poor quality of life. The characteristics are close to European studies

Natural evolution can lead to a total physical, psychological, social deconditioning. A link has been established between the severity of this pathology, a provider of precariousness and the poor physical condition, related to physical inactivity. The reverse has been described , so the practice of APA brings a significant reduction in symptoms .

To our knowledge, no study has demonstrated with sufficient evidence the effectiveness of the practice of well-defined adapted physical activity (APA) via a reproducible program of physical activity that has been the mechanisms of action that underlie this efficacy by biology and functional brain imaging (PET CT) in this context.

In addition, the publications mention recruitment difficulties, a high drop-out rate and a difficult maintenance of the benefits of physical activity in the long term, or even a return to the initial level after a few months.

The programs evaluated do not seem to take into account the peculiarities of patients, their coping coping strategies, associated with chronic pain and disability . In order to reinforce the durability of the benefits of our intervention, we make modulating factors of "coping" styles of therapeutic targets in their own right, as well as muscular strength, aerobic capacity or flexibility. Thus, cognitive-behavioral therapy (CBT) procedures validated in the treatment of chronic pain are adapted and transposed to our APA program in order to propose specific strategies.

"Fibromy'activ" aims to act upstream and downstream of the formation of health inequalities found in the population suffering from fibromyalgia and favored by the natural evolution of the disease: These workshops tend to favorably influence the course of life and to define a reproducible interdisciplinary protocol.

It is a question of making accessible and reproducible the practice of adapted physical activity (APA), non-medicinal therapeutic recommended by the HAS since 2010 (level of proof A), by the EULAR in 2016, but not refunded, poorly protocolized therefore not reproducible and little implementation. It is part of the spirit of the amended Health Act with the coming into force of the application decree since March 2017 "Physical Prescription".

ELIGIBILITY:
Inclusion Criteria:

Female or male subject, 18 years of age or older, not pregnant, not breastfeeding, not deprived of liberty;

* Subject with fibromyalgia meeting the criteria of the American College of Rheumatology (ACR)
* Subject managed by the Center for Assessment and Pain Management of CHU Timone or addressed to it in consultation / day hospital;
* Subject free from any general illness or serious psychiatric disorders, and any infectious, inflammatory, tumoral, vascular, degenerative or traumatic pathology of the central nervous system, determined during the interrogation;
* Subject not having a history of alcoholism or drug addiction,
* Subject with no contraindication to PET scintigraphy (pregnancy and lactation),
* Subject with no indication of physical activity;
* Subject whose general state and comprehension of French makes it possible to complete a questionnaire;
* Topic with average pain> 4/10 at EN
* Subject affiliated with Social Security
* Subject who has read, understood and signed informed consent after informing and accepting protocol rules

Exclusion Criteria:

• Major subject under legal protection or unable to express their consent: L1121-8 of the CSP

* Subject presenting a contraindication to the practice of physical activity, to scintigraphic scanning by PET,
* Subject deprived of liberty following a judicial or administrative decision
* Subject with psychiatric illness or Personality Disorder making group work difficult
* Subject refusing to participate in the study or not signing the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire | 1 hour
  FIQ Questionnaire was developed in 1991 as a specific measuring instrument for assessing the health status of patients with fibromyalgia. The validation of this adaptation and the evaluation of its psychometric properties were carried out by Perrot in 2002.
  self-administered, exploring ten dimensions of the impact of pathology on quality of life.
  Scale from 0 to 10, a high figure corresponding to a greater disadvantage or handicap. The analysis of the evolution of the FIQ over time, spontaneously or under treatment, is therefore dimension by dimension, in order to maintain a clinical informative value, as well as by an aggregate score ( corresponding to the algebraic sum of the dimensions evaluated, compared to 100 units). A weighting of the aggregate score is expected when the patient can not assess impact on professional activity.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France